CLINICAL TRIAL: NCT02078674
Title: A Phase I/II Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of Monovalent A/Anhui/1/13 (H7N9) Virus-Like Particle (VLP) Avian Influenza Antigen (Recombinant) in Healthy Adults With and Without Matrix-M1™
Brief Title: A(H7N9) VLP Antigen Dose-Ranging Study With Matrix-M1™ Adjuvant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FLU-MI7A-201
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Influenza (Pandemic)
Keywords: H7N9
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group A (Experimental): Placebo
  Interventions: Biological: Placebo
- Group B (Experimental): High dose Monovalent Avian Influenza VLP (H7N9); IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9)
- Group C (Experimental): High dose Monovalent Avian Influenza VLP (H7N9) with Low dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant
- Group D (Experimental): Intermediate dose Monovalent Avian Influenza VLP (H7N9) with Low dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant
- Group E (Experimental): Low dose Monovalent Avian Influenza VLP (H7N9) with Low dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant
- Group F (Experimental): High dose Monovalent Avian Influenza VLP (H7N9) with High dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant
- Group G (Experimental): Intermediate dose Monovalent Avian Influenza VLP (H7N9) with High dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant
- Group H (Experimental): Low dose Monovalent Avian Influenza VLP (H7N9) with High dose Matrix-M1™ adjuvant; IM; Day 0 and Day 21
  Interventions: Biological: Monovalent Avian Influenza VLP (H7N9); Biological: Matrix-M1™ adjuvant

INTERVENTIONS:
Biological: Monovalent Avian Influenza VLP (H7N9)
  Arms: Group B; Group C; Group D; Group E; Group F; Group G; Group H
Biological: Matrix-M1™ adjuvant
  Arms: Group C; Group D; Group E; Group F; Group G; Group H
Biological: Placebo
  Arms: Group A

SUMMARY:
This is a randomized, observer-blinded, placebo-controlled trial in adults 18 to 64 years old. Randomization will be stratified by age (18 to 49 years and 50 to 64 years) and by prior influenza immunization within the past three months. Subjects 18 to 49 years of age will comprise ~67% of subjects in each treatment group, and the balance will comprise subjects 50 to 64 years.

Each subject will receive two identical IM doses of test article at a 21-day interval (Day 0 and Day 21), in alternate deltoids. For each subject, study follow-up will span approximately 385 days total, or approximately 13 months from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female, 18 to 64 years of age,
2. Willing and able to give informed consent prior to study enrollment,
3. Able to comply with study requirements, and
4. Women of child-bearing potential must have a negative urine pregnancy test prior to each vaccination, and will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of continuous abstinence from heterosexual activity or prior surgical sterilization, hormonal contraceptives (oral, injectable, implant, patch, ring), barrier contraceptives (condom or diaphragm), and intrauterine device (IUD). Women with an adequately documented history of surgical sterility, or ≥50 years of age and without menses for ≥1 year are exempt from urine pregnancy testing.

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care.

   * Asymptomatic conditions or findings (e.g., mild hypertension, dyslipidemia) that are not associated with evidence of end-organ damage are not exclusionary provided that they are being appropriately managed and are clinically stable (i.e., unlikely to result in symptomatic illness within the time-course of this study) in the opinion of the Investigator.
   * Acute or chronic illnesses or conditions which may be reasonably predicted to become symptomatic if treatment were withdrawn or interrupted are exclusionary, even if stable.
   * Note that illnesses or conditions may be exclusionary, even if otherwise stable and clinically minor, due to therapies used to treat them (see exclusion criteria 3, 5, 8, 9).
2. Any grade 1 or higher (as based on the Toxicity Grading Scale [TGS]) abnormality in ALT, AST, alkaline phosphatase, total bilirubin, blood urea nitrogen, or creatinine levels.
3. Any grade 2 or higher (as based on the TGS) vital sign or clinical laboratory abnormality not specified in criterion 2 above. Note that any abnormal vital sign may be repeated at the Investigator's discretion.
4. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
5. History of a serious reaction to prior influenza vaccination.
6. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
7. Received any vaccine in the 4 weeks preceding the study vaccination; or any A(H7N9) avian influenza vaccine at any time.
8. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
9. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
10. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
11. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
12. Known disturbance of coagulation.
13. Women who are pregnant or breastfeeding, or plan to become pregnant during the study.
14. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 610 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Assessment of Safety | Day 0 to Day 384
  Counts (and percentages) of subjects with solicited local and systemic AEs over the seven days post-injection and all adverse events, solicited and unsolicited, including adverse changes in clinical laboratory parameters, over 42 days post-first injection.
  In addition, MAEs, SAEs, and SNMCs will be collected for one year.
Immunogenicity as assessed by hemagglutination-inhibiting (HAI) antibody titers against the vaccine-homologous A/Anhui/1/13 (H7N9) virus. | Day 0 to Day 384
  Geometric mean titer (GMT) Geometric mean ratio (GMR) Seroconversion rate (SCR) Seroresponse rate (SRR)

SECONDARY OUTCOMES:
Immunogenicity as assessed by neuraminidase-inhibiting antibodies to N9. | Day 0 to Day 384

CONTACTS AND LOCATIONS:
Overall Officials: D. Nigel Thomas, Ph. D., Study Director — Novavax, Inc.
Locations (5):
- United States (5):
  - Diablo Clinical Research, Walnut Creek, California
  - Miami Research Associates, Miami, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Regional Clinical Research, Inc., Endwell, New York
  - Coastal Carolina Research, Mt. Pleasant, South Carolina